CLINICAL TRIAL: NCT01094288
Title: A Phase 1 Study of MLN8237, an Aurora A Kinase Inhibitor, in Patients With Advanced Solid Tumors Including Castration-Resistant Prostate Cancer Receiving a Standard Docetaxel Regimen
Brief Title: A Phase 1 Study of Alisertib Participants With Advanced Solid Tumors Including Castration-Resistant Prostate Cancer Receiving a Standard Docetaxel Regimen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C14009
Record Dates: First submitted 2010-03-17; First posted 2010-03-26 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-10

CONDITIONS: Advanced Solid Tumors; Adenocarcinoma of the Prostate
MeSH Terms: interventions — MLN 8237; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Alisertib + Docetaxel (Experimental): Alisertib in escalating dose (10-40 mg), enteric-coated tablets (ECT), orally, twice daily for 7 days followed by 14-day rest period in Cycle 1, 3 and onwards (21-day cycle) and orally twice daily from Day 3 to Day 7 followed by 14 day rest period in Cycle 2 along with docetaxel 60-75 mg/m^2, intravenous (IV) infusion on Day 1 of each cycle for maximum of 12 months, or until the occurrence of progressive disease (PD), unmanageable adverse events (AEs) or withdrawal of consent.
  The starting alisertib dose is 10 mg, orally, twice daily (total 20 mg/day).
  Interventions: Drug: Alisertib; Drug: Docetaxel

INTERVENTIONS:
Drug: Alisertib — Alisertib ECT
  Other Names: MLN8237
Drug: Docetaxel — Docetaxel IV infusion

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of alisertib in combination with docetaxel as a treatment for participants with advanced solid tumors, including castration-resistant prostate cancer, who were deemed by the investigator to be medically appropriate candidates for docetaxel therapy.

DETAILED DESCRIPTION:
The drug being tested in this study is called alisertib (MLN8237). Alisertib is being tested to treat people who have advanced solid tumors including castration-resistant prostate cancer.

The study enrolled approximately 41 patients. Participants were enrolled to receive:

• Alisertib 10-40 mg + docetaxel 60-75 mg/m^2

All participants will receive alisertib (ECT) in dose escalating cohorts, orally, twice daily for 7 days followed by 14-day rest period in Cycle 1, 3 and onwards (21-day cycle) and orally twice daily from Day 3 to Day 7 followed by 14 day rest period in Cycle 2 [dose held for pharmacokinetic (PK) collection] along with docetaxel 75 mg/m^2, intravenous (IV) infusion on Day 1 of each cycle for maximum of 12 months, or until the occurrence of progressive disease (PD), unmanageable AEs or withdrawal of consent.

This multi-center trial is conducted in United States. The overall time to participate in this study was until there is evidence of disease progression or unacceptable treatment-related toxicity. Participants made multiple visits to the clinic, and were contacted every 12 weeks for up to 25.8 months after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

Each participant must meet all of the following inclusion criteria to be enrolled in the study:

* 18 years or older
* Histologically or cytologically confirmed advanced tumors and candidates for docetaxel treatment
* Measurable or evaluable disease is required. Participants must have clinical evidence of progressive disease or persistent disease
* Participants with castration-resistant prostate cancer (CRPC) are required to have

  * Pathologically confirmed adenocarcinoma of the prostate
  * Evidence of metastatic disease on bone scan or other imaging. Participants with prostate-specific antigen (PSA) elevation as the only manifestation of disease are not eligible.
  * Progressive disease after at least 1 hormonal treatment with documented testosterone levels less than 50 ng/dl
  * Concurrent use of an agent for testosterone suppression (e.g., luteinizing hormone-releasing hormone [LHRH] agonist) is required if the participants has not been surgically castrated
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Recovered to less than or equal to Grade 1 toxicity (CTCAE), to participant's baseline status (except alopecia) or deemed irreversible from the effects of prior cancer therapy and must have evidence of progressive or persistent disease
* Adequate bone marrow, liver and renal function
* Any use of opiates must be stable for at least 2 weeks prior to study entry
* Female participants who are postmenopausal for at least 1 year OR are surgically sterile OR if of childbearing potential, agree to practice 2 effective methods of contraception at the same time
* Male participants who agree to practice effective barrier contraception during the entire study and through 6 months after the last dose of study drug OR agree to abstain from heterosexual intercourse
* Voluntary written consent
* Willing to comply with scheduled visits, treatment plan, laboratory tests and other trial procedures
* Suitable venous access for blood sampling

Exclusion Criteria:

Participants meeting any of the following exclusion criteria are not to be enrolled in the study:

* Female participants who are lactating or pregnant
* Antineoplastic therapy or any experimental therapy within 21 days before the first dose of alisertib
* Prior or current investigational therapies within 4 weeks before the first dose of MLN8237
* Concurrent investigational treatment of treatment with any investigational products within 28 days before the first dose of alisertib
* Radiotherapy to greater than 40% of bone marrow or any radiotherapy (except localized, small field radiation) within 4 weeks prior to enrollment, unless reviewed and approved by the medical monitor
* Nitrosoureas or mitomycin-C within 6 weeks before the first dose of alisertib.
* Autologous stem cell transplant within 3 months before the first dose of alisetib, or prior allogeneic stem cell transplant at any time.
* Use of enzyme-inducing antiepileptic drugs such as phenytoin, carbamazepine or phenobarbital, or rifampin, rifabutin, rifapentine or St. John's wort within 14 days prior to the first dose of alisertib
* For CRPC participants:

  * Radiotherapy or antiandrogen therapy for prostate cancer within 4 weeks prior to enrollment
  * Prior treatment with antineoplastic chemotherapy or radioisotopes for advanced prostate cancer
  * Use of products known to affect PSA levels within 4 weeks of enrollment
* Major surgery within 4 weeks of study enrollment
* Uncontrolled high blood pressure
* Participants with abnormal gastric or bowel function or who require continuous treatment with antacids or proton pump inhibitors
* Participants receiving chronic steroid therapy other than the following: low dose steroid for the control of nausea and vomiting, topical steroid, inhaled steroid or use of dexamethasone
* Known severe hypersensitivity to docetaxel or other drugs formulated in polysorbate 80
* Comorbid condition or unresolved toxicity that would preclude administration of docetaxel
* Prior history of Grade 2 or greater neurotoxicity or any toxicity that has not resolved to Grade 1 or below
* Symptomatic brain or other CNS metastasis
* Diagnosis or treatment of another malignancy within 2 years preceding first dose of study drug except nonmelanoma skin cancer or in situ malignancy completely resected
* Known history of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C
* Participants requiring full systemic anticoagulation
* Prior allogeneic bone marrow or other organ transplant
* Active infection requiring systemic therapy within 14 days preceding first dose, or other serious infection
* History of hemorrhagic or thrombotic cerebrovascular event in the past 12 months
* Serious medical or psychiatric illness that could interfere with protocol completion
* Inability to swallow oral medication
* Prior treatment with more than 3 myelosuppressive cytotoxic chemotherapy regimens
* Prior treatment with more than 1 prior taxane-containing regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-08-17 (Actual); Primary Completion 2014-02-28 (Actual); Study Completion 2017-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (4):
- United States (4):
  - Indianapolis, Indiana
  - Portland, Oregon
  - San Antonio, Texas
  - Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 investigative sites in the United States from 17 August 2010 to 04 January 2017.
Pre-assignment Details: Participants with a diagnosis of Advanced solid tumors, including castration-resistant prostate cancer were enrolled to receive alisertib Alisertib 10-40 mg + docetaxel 60-75 mg/m^2 intravenous (IV) infusion and granulocyte colony stimulating factor (GCSF) in escalating dose cohorts.
Groups:
- Alisertib 10 mg (7D) + Docetaxel 75 mg/m^2: Alisertib 10 mg, enteric-coated tablets (ECT), orally, twice daily for 7 days in Cycle 1, 3 and onwards; and orally twice daily from Day 3 to Day 7 in Cycle 2 followed by 14 day rest period along with docetaxel 75 mg/m^2, intravenous infusion on Day 1 of each cycle (21-day cycle) for a maximum of 28 cycles, or until the occurrence of PD, unmanageable adverse events (AEs) or withdrawal of consent.
- Alisertib 20 mg (7D) + Docetaxel 75 mg/m^2: Alisertib 20 mg, ECT, orally, twice daily for 7 days in Cycle 1, 3 and onwards; and orally twice daily from Day 3 to Day 7 in Cycle 2 followed by 14 day rest period along with docetaxel 75 mg/m^2, intravenous infusion on Day 1 of each cycle (21-day cycle) for a maximum of 34 cycles, or until the occurrence of PD, unmanageable AEs or withdrawal of consent.
- Alisertib 30 mg (7D) + Docetaxel 75 mg/m^2: Alisertib 30 mg, ECT, orally, twice daily for 7 days in Cycle 1, 3 and onwards; and orally twice daily from Day 3 to Day 7 in Cycle 2 followed by 14 day rest period along with docetaxel 75 mg/m^2, intravenous infusion on Day 1 of each cycle (21-day cycle) for a maximum of 36 cycles, or until the occurrence of PD, unmanageable AEs or withdrawal of consent.
- Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2: Alisertib 30 mg, ECT, orally, twice daily for 5 days in Cycle 1, 3 and onwards; and orally twice daily from Day 3 to Day 7 in Cycle 2 followed by 14 day rest period along with docetaxel 75 mg/m^2, intravenous infusion on Day 1 of each cycle (21-day cycle) for a maximum of 17 cycles, or until the occurrence of PD, unmanageable AEs or withdrawal of consent.
- Alisertib 30 mg (7D) + Docetaxel 60 mg/m^2: Alisertib 30 mg, ECT, orally, twice daily for 7 days in Cycle 1, 3 and onwards; and orally twice daily from Day 3 to Day 7 in Cycle 2 followed by 14 day rest period along with docetaxel 60 mg/m^2, intravenous infusion on Day 1 of each cycle (21-day cycle) for a maximum of 15 cycles, or until the occurrence of PD, unmanageable AEs or withdrawal of consent.
- Alisertib 30 mg (5D) + Docetaxel 60 mg/m^2: Alisertib 30 mg, ECT, orally, twice daily for 5 days in Cycle 1, 3 and onwards; and orally twice daily from Day 3 to Day 7 in Cycle 2 followed by 14 day rest period along with docetaxel 60 mg/m^2, intravenous infusion on Day 1 of each cycle (21-day cycle) for a maximum of 5 cycles, or until the occurrence of PD, unmanageable AEs or withdrawal of consent.
- Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 + GCSF: Alisertib 30 mg, ECT, orally, twice daily for 5 days in Cycle 1, 3 and onwards; and orally twice daily from Day 3 to Day 7 in Cycle 2 followed by 14 day rest period along with docetaxel 75 mg/m^2, intravenous infusion on Day 1 of each cycle (21-day cycle) and granulocyte colony stimulating factor (GCSF) as per standard of care for a maximum of 2 cycles, or until the occurrence of PD, unmanageable AEs or withdrawal of consent.
- Alisertib 40 mg (5D) + Docetaxel 75 mg/m^2 + GCSF: Alisertib 40 mg, ECT, orally, twice daily for 5 days in Cycle 1, 3 and onwards; and orally twice daily from Day 3 to Day 7 in Cycle 2 followed by 14 day rest period along with docetaxel 75 mg/m^2, intravenous infusion on Day 1 of each cycle (21-day cycle) and granulocyte colony stimulating factor (GCSF) as per standard of care for a maximum of 5 cycles, or until the occurrence of PD, unmanageable AEs or withdrawal of consent.
Period: Overall Study
Arm/Group | Alisertib 10 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 20 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 + GCSF | Alisertib 40 mg (5D) + Docetaxel 75 mg/m^2 + GCSF
Started | 6 | 15 | 5 | 3 | 2 | 4 | 2 | 4
Completed | 4 (Completed=Completed Treatment) | 5 | 1 | 1 | 2 | 4 | 2 | 2
Not Completed | 2 | 10 | 4 | 2 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2
Not completed — Initiation of Alternative Therapy | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Reason not Specified | 2 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Ongoing Participants | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received at least 1 dose of any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Alisertib 10 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 20 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 + GCSF | Alisertib 40 mg (5D) + Docetaxel 75 mg/m^2 + GCSF | Total
Number analyzed (Participants) | 6 | 15 | 5 | 3 | 2 | 4 | 2 | 4 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (5.20) | 61.5 (13.10) | 60.2 (16.75) | 61.3 (8.62) | 56.5 (2.12) | 54.8 (18.73) | 52.5 (26.16) | 62.3 (25.71) | 60.4 (14.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 1 | 1 | 1 | 1 | 2 | 1 | 11
  Male | 6 | 11 | 4 | 2 | 1 | 3 | 0 | 3 | 30
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 0 | 5 | 0 | 0 | 0 | 1 | 1 | 0 | 7
  Not Hispanic or Latino | 6 | 10 | 5 | 3 | 1 | 3 | 1 | 4 | 33
  Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  White | 6 | 15 | 5 | 2 | 2 | 3 | 2 | 3 | 38
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Other | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 15 | 5 | 3 | 2 | 4 | 2 | 4 | 41
Height [Mean (Standard Deviation); unit: cm] | 185.5 (11.02) | 170.5 (10.04) | 177.2 (12.13) | 171.0 (10.08) | 174.5 (0.71) | 172.5 (10.98) | 155.6 (8.08) | 174.9 (6.99) | 173.6 (11.32)
Weight [Mean (Standard Deviation); unit: kg] | 100.25 (15.842) | 82.73 (16.963) | 94.15 (25.623) | 87.73 (31.987) | 76.90 (8.344) | 85.97 (15.987) | 62.05 (11.950) | 87.05 (21.025) | 86.50 (19.550)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] — BSA (m^2) = square root [height (cm) * weight (kg)/3600].
  m^2 | 2.269 (0.2329) | 1.973 (0.2533) | 2.138 (0.3541) | 2.025 (0.4316) | 1.929 (0.1009) | 2.026 (0.2420) | 1.635 (0.2005) | 2.046 (0.2945) | 2.034 (0.2878)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study were reported as adverse events. A SAE is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: From enrollment through 30 days after the last dose of study drug (approximately up to 77 months)
Population: Safety Population included all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Alisertib 10 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 20 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 + GCSF | Alisertib 40 mg (5D) + Docetaxel 75 mg/m^2 + GCSF
Number analyzed (Participants) | 6 | 15 | 5 | 3 | 2 | 4 | 2 | 4
participants
  AEs | 6 | 15 | 5 | 3 | 2 | 4 | 2 | 4
  SAEs | 3 | 8 | 3 | 2 | 1 | 3 | 2 | 2

2. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Docetaxel
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose in Cycles 1 and 2
Population: Pharmacokinetic (PK) parameter population was defined as all participants who had sufficient dosing data and plasma alisertib or docetaxel concentration-time data to permit the calculation of any PK parameter. Here number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Alisertib 10 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 20 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 + GCSF | Alisertib 40 mg (5D) + Docetaxel 75 mg/m^2 + GCSF
Number analyzed (Participants) | 6 | 15 | 5 | 3 | 2 | 4 | 2 | 4
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 6 | 13 | 5 | 3 | 2 | 4 | 2 | 4
  Cycle 1 Day 1 | 2392.7 (60.2) | 1730.4 (26.5) | 1587.0 (34.1) | 1717.6 (51.9) | 3751.4 (80.8) | 1159.9 (13.8) | 2232.9 (19.8) | 1386.6 (47.0)
  Cycle 2 Day 1: number analyzed (Participants) | 6 | 9 | 4 | 2 | 2 | 4 | 2 | 2
  Cycle 2 Day 1 | 1825.1 (25.9) | 1957.0 (23.4) | 2146.6 (19.4) | 3299.9 (0.9) | 1649.7 (19.1) | 1061.6 (24.8) | 2504.6 (28.0) | 1627.8 (17.2)

3. Secondary Outcome: AUC(Last): Area Under the Plasma Concentration Curve From Time 0 to the Time of the Last Quantifiable Concentration for Docetaxel
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose in Cycles 1 and 2
Population: PK parameter population was defined as all participants who had sufficient dosing data and plasma alisertib or docetaxel concentration-time data to permit the calculation of any PK parameter. Here number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Alisertib 10 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 20 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 + GCSF | Alisertib 40 mg (5D) + Docetaxel 75 mg/m^2 + GCSF
Number analyzed (Participants) | 6 | 15 | 5 | 3 | 2 | 4 | 2 | 4
hr*ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 6 | 13 | 4 | 3 | 1 | 3 | 2 | 4
  Cycle 1 Day 1 | 2328.3 (69.5) | 1925.7 (21.4) | 1750.1 (23.1) | 2163.4 (52.8) | 1830.0 (NA) — Geometric coefficient of variation is not estimable as only 1 participants is assessed. | 1593.1 (14.0) | 2394.6 (2.7) | 1579.8 (45.4)
  Cycle 2 Day 1: number analyzed (Participants) | 5 | 9 | 3 | 2 | 2 | 3 | 2 | 1
  Cycle 2 Day 1 | 1750.8 (23.1) | 2416.4 (23.7) | 25.5 (2174.6) | 7811.5 (87.5) | 1622.8 (35.0) | 1596.0 (19.9) | 2895.7 (16.3) | 2510.0 (NA) — Geometric coefficient of variation is not estimable as only 1 participants is assessed.

4. Secondary Outcome: AUC∞: Area Under the Plasma Concentration Curve From Time 0 to Infinity for Docetaxel
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose in Cycles 1 and 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Alisertib 10 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 20 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 + GCSF | Alisertib 40 mg (5D) + Docetaxel 75 mg/m^2 + GCSF
Number analyzed (Participants) | 6 | 15 | 5 | 3 | 2 | 4 | 2 | 4
hr*ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 5 | 9 | 4 | 1 | 1 | 3 | 2 | 3
  Cycle 1 Day 1 | 2653.3 (68.1) | 2240.6 (23.9) | 2007.3 (15.7) | 3570.0 (NA) — Geometric Coefficient of Variation is not estimable as only 1 participants is assessed. | 2130.0 (NA) — Geometric Coefficient of Variation is not estimable as only 1 participants is assessed. | 1734.7 (9.6) | 2600.0 (0.0) | 1730.9 (53.9)
  Cycle 2 Day 1: number analyzed (Participants) | 5 | 8 | 2 | 1 | 2 | 2 | 2 | 1
  Cycle 2 Day 1 | 1918.0 (21.4) | 2632.2 (28.0) | 2019.8 (10.1) | 4000.0 (NA) — Geometric Coefficient of Variation is not estimable as only 1 participants is assessed. | 1785.4 (35.6) | 1631.0 (9.9) | 3099.0 (14.3) | 3120.0 (NA) — Geometric Coefficient of Variation is not estimable as only 1 participants is assessed.

5. Secondary Outcome: Terminal Phase Elimination Half-life (T1/2) for Docetaxel
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose in Cycles 1 and 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Alisertib 10 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 20 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 + GCSF | Alisertib 40 mg (5D) + Docetaxel 75 mg/m^2 + GCSF
Number analyzed (Participants) | 6 | 15 | 5 | 3 | 2 | 4 | 2 | 4
hr
  Cycle 1 Day 1: number analyzed (Participants) | 5 | 9 | 4 | 1 | 1 | 3 | 2 | 3
  Cycle 1 Day 1 | 21.80 (4.339) | 22.88 (4.733) | 24.00 (6.934) | 15.60 (NA) — Standard deviation is not estimable as only 1 participants is assessed. | 30.70 (NA) — Standard deviation is not estimable as only 1 participants is assessed. | 16.34 (5.684) | 19.25 (2.051) | 24.80 (6.444)
  Cycle 2 Day 1: number analyzed (Participants) | 5 | 8 | 2 | 1 | 2 | 2 | 2 | 1
  Cycle 2 Day 1 | 24.18 (2.050) | 20.73 (5.845) | 20.40 (2.121) | 16.40 (NA) — Standard deviation is not estimable as only 1 participants is assessed. | 25.10 (2.546) | 22.00 (2.404) | 16.95 (0.636) | 26.00 (NA) — Standard deviation is not estimable as only 1 participants is assessed.

6. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Alisertib
Time Frame: Prior to dosing on Day 1 and Day 5 or 7 and at multiple time points (up to 12 hours) post-dose in Cycle 1
Population: PK parameter population was defined as all participants who had sufficient dosing data and plasma alisertib concentration-time data to permit the calculation of any PK parameter. Here number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- Alisertib 10 mg: Alisertib 10 mg, ECT, orally, twice daily for 7 days in Cycle 1, 3 and onwards; and orally twice daily from Day 3 to Day 7 in Cycle 2 of each cycle (21-day cycle).
- Alisertib 20 mg: Alisertib 20 mg, ECT, orally, twice daily for 7 days in Cycle 1, 3 and onwards; and orally twice daily from Day 3 to Day 7 in Cycle 2.
- Alisertib 30 mg: Alisertib 30 mg, ECT, orally, twice daily for 7 days in Cycle 1, 3 and onwards; and orally twice daily from Day 3 to Day 7 in Cycle 2. Assessment was performed on Day 5 if alisertib was given on a 5 day schedule.
- Alisertib 40 mg: Alisertib 40 mg, ECT, orally, twice daily for 7 days in Cycle 1, 3 and onwards; and orally twice daily from Day 3 to Day 7 in Cycle 2. Assessment was performed on Day 5 if alisertib was given on a 5 day schedule.
Arm/Group | Alisertib 10 mg | Alisertib 20 mg | Alisertib 30 mg | Alisertib 40 mg
Number analyzed (Participants) | 6 | 15 | 16 | 4
nmol/L
  Cycle 1 Day 1: number analyzed (Participants) | 5 | 15 | 16 | 4
  Cycle 1 Day 1 | 290.4 (22.1) | 557.5 (57.3) | 751.6 (31.3) | 1346.4 (49.8)
  Cycle 1 Day 5/Day 7: number analyzed (Participants) | 6 | 13 | 11 | 4
  Cycle 1 Day 5/Day 7 | 435.8 (31.0) | 1140.6 (44.7) | 1637.9 (52.1) | 1766.3 (40.1)

7. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Alisertib
Time Frame: Prior to dosing on Day 1 and Day 5 or 7 and at multiple time points (up to 12 hours) post-dose in Cycle 1
Population: as for outcome 6
Measure: Median (Full Range); unit: hr
Arm/Group | Alisertib 10 mg | Alisertib 20 mg | Alisertib 30 mg | Alisertib 40 mg
Number analyzed (Participants) | 6 | 15 | 26 | 4
hr
  Cycle 1 Day 1: number analyzed (Participants) | 5 | 15 | 16 | 4
  Cycle 1 Day 1 | 2.050 [2.00 to 3.00] | 4.000 [2.00 to 9.98] | 3.560 [2.00 to 12.00] | 1.500 [1.00 to 7.58]
  Cycle 1 Day 5/Day 7: number analyzed (Participants) | 6 | 13 | 11 | 4
  Cycle 1 Day 5/Day 7 | 3.510 [1.87 to 8.22] | 3.030 [2.00 to 9.40] | 2.030 [2.00 to 8.00] | 1.975 [1.08 to 3.00]

8. Secondary Outcome: AUCτ: Area Under the Plasma Concentration-time Curve From Time 0 to Day 7 Over the Dosing Interval for Alisertib
Time Frame: Prior to dosing on Day 1 and Day 5 or 7 and at multiple time points (up to 12 hours) post-dose in Cycle 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nmol/L
Arm/Group | Alisertib 10 mg | Alisertib 20 mg | Alisertib 30 mg | Alisertib 40 mg
Number analyzed (Participants) | 6 | 15 | 16 | 4
hr*nmol/L
  Cycle 1 Day 1: number analyzed (Participants) | 5 | 15 | 16 | 4
  Cycle 1 Day 1 | 1635.0 (28.3) | 3303.0 (46.1) | 4387.5 (30.1) | 8013.7 (43.1)
  Cycle 1 Day 5/Day 7: number analyzed (Participants) | 6 | 13 | 11 | 4
  Cycle 1 Day 5/Day 7 | 3052.8 (42.0) | 8546.0 (49.7) | 13199.1 (60.8) | 12630.0 (27.7)

9. Secondary Outcome: Overall Response Rate (ORR) Assessed for Overall Participant Population
Description: ORR is defined as percentage of participants who achieved complete response (CR) or partial response (PR) as assessed by response evaluation criteria in solid tumors (RECIST) v 1.1. CR was defined as disappearance of all target and non-target lesions and normalization of tumor marker levels. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as ≥30% decrease in sum of longest diameter (LD) of target lesions in reference to Baseline. RECIST-Evaluable Population is subset of safety population who had measurable disease by RECIST v 1.1 at baseline and had at least 1 post baseline response. prostate specific antigen (PSA)-Evaluable Population is subset of the safety population who had a baseline PSA reference value (>5 ng/mL) and at least 12 weeks post-baseline PSA assessment for participants with no decline from baseline, or PSA progression within 12 weeks of treatment for participants with PSA decline from baseline.
Time Frame: Baseline up to Cycle 36 (21-day cycles) until disease progression, death or EOT (approximately up to 24.8 months)
Population: Response-Evaluable Population included participants who were either RECIST evaluable and/or PSA-evaluable.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alisertib 10 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 20 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 + GCSF | Alisertib 40 mg (5D) + Docetaxel 75 mg/m^2 + GCSF
Number analyzed (Participants) | 6 | 10 | 1 | 2 | 2 | 4 | 1 | 2
percentage of participants | 50 [12 to 88] | 10 [0 to 45] | 100 [NA to NA] — 95% Confidence Interval is not estimable as only 1 participants is assessed. | 50 [1 to 99] | 0 [0 to 0] | 25 [1 to 81] | 0 [0 to 0] | 50 [1 to 99]

10. Secondary Outcome: Overall Response Rate for Prostate Cancer Participants
Description: ORR is defined as percentage of participants who achieved CR or PR as assessed by either RECIST v 1.1 or PSA response by prostate cancer working group 2 (PCWG2) criteria. According to RECIST v 1.1, CR: disappearance of all target and non-target lesions and (if applicable) normalization of tumor marker levels. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: ≥30% decrease in sum of LD of target lesions in reference to Baseline sum LD. PSA response by PCWG2 is defined as PSA at least 50% decrease in PSA value from baseline for 2 consecutive evaluations. PCWG2 defines PSA progression as the date that a 25% or greater increase and an absolute increase of 2 ng/mL or more from the nadir is documented, which is confirmed by a second value obtained 3 or more weeks later.
Time Frame: Baseline up to Cycle 36 (21-day cycles) until disease progression, death or EOT (approximately up to 24.8 months)
Population: Response-Evaluable Population included participants who were either RECIST evaluable or PSA-evaluable. Here, number of participants analyzed are the enrolled participants who had castration-resistant prostate cancer (CRPC) and were evaluable by either RECIST or PSA response criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alisertib 10 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 20 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 + GCSF | Alisertib 40 mg (5D) + Docetaxel 75 mg/m^2 + GCSF
Number analyzed (Participants) | 6 | 5 | 0 | 1 | 0 | 1 | 0 | 1
percentage of participants | 50 [12 to 88] | 20 [1 to 72] |  | 100 [NA to NA] — 95% Confidence Interval is not estimable as only 1 participants is assessed. |  | 0 [0 to 0] |  | 100 [NA to NA] — 95% Confidence Interval is not estimable as only 1 participants is assessed.

11. Secondary Outcome: Best Overall Response Rate Assessed by RECIST Criteria
Description: Best response rate is defined as the percentage of participants with CR, PR, CR+PR, stable disease (SD) and progressive disease (PD) as assessed by RECIST criteria 1.1 for target lesions and assessed by CT, PET or MRI. CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: Baseline up to Cycle 36 (21-day cycles) until disease progression, death or EOT (approximately up to 24.8 months)
Population: RECIST-Evaluable Population included a subset of the safety population who had measurable disease by RECIST v 1.1 at baseline and had at least 1 post baseline response assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alisertib 10 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 20 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 + GCSF | Alisertib 40 mg (5D) + Docetaxel 75 mg/m^2 + GCSF
Number analyzed (Participants) | 6 | 9 | 1 | 2 | 2 | 4 | 1 | 2
percentage of participants
  Complete Response (CR) | 0 [0 to 0] | 0 [0 to 0] | 100 [NA to NA] — 95% Confidence Interval is not estimable as only 1 participants is assessed. | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Partial Response (PR) | 50 [12 to 88] | 11 [0 to 48] | 0 [0 to 0] | 50 [1 to 99] | 0 [0 to 0] | 25 [1 to 81] | 0 [0 to 0] | 50 [1 to 99]
  CR+PR | 50 [12 to 88] | 11 [0 to 48] | 100 [NA to NA] — 95% Confidence Interval is not estimable as only 1 participants is assessed. | 50 [1 to 99] | 0 [0 to 0] | 25 [1 to 81] | 0 [0 to 0] | 50 [1 to 99]
  Stable Disease (SD) | 50 [12 to 88] | 67 [30 to 93] | 0 [0 to 0] | 0 [0 to 0] | 50 [1 to 99] | 0 [0 to 0] | 0 [0 to 0] | 50 [1 to 99]
  Progressive Disease (PD) | 0 [0 to 0] | 22 [3 to 60] | 0 [0 to 0] | 50 [1 to 99] | 50 [1 to 99] | 75 [19 to 99] | 100 [NA to NA] — 95% Confidence Interval is not estimable as only 1 participants is assessed. | 0 [0 to 0]

12. Secondary Outcome: Best Overall Response Rate Assessed by PSA Response by Prostate Cancer Working Group 2 (PCWG2) Criteria
Description: Best Response Assessed by PSA Response by Prostate Cancer Working Group 2 (PCWG2) Criteria PSA response is defined as at least 50% decrease in PSA value from baseline for 2 consecutive evaluations.
Time Frame: Baseline up to Cycle 36 (21-day cycles) until disease progression, death or EOT (approximately up to 24.8 months)
Population: PSA-Evaluable Population is a subset of the safety population who had a baseline PSA reference value (>5 ng/mL) and at least 12 weeks post-baseline PSA assessment for participants with no decline from baseline, or PSA progression within 12 weeks of treatment for participants with PSA decline from baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alisertib 10 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 20 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 + GCSF | Alisertib 40 mg (5D) + Docetaxel 75 mg/m^2 + GCSF
Number analyzed (Participants) | 6 | 5 | 0 | 1 | 0 | 0 | 0 | 0
percentage of participants
  ≥50% Reduction from Baseline | 67 [22 to 96] | 80 [28 to 99] |  | 100 [NA to NA] — 95% Confidence Interval is not estimable as only 1 participants is assessed. |  |  |  |
  <50% Reduction from Baseline | 33 [4 to 78] | 20 [1 to 72] |  | 0 [0 to 0] |  |  |  |

13. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from the date of first documentation of a response to the date of first documented progressive disease (PD), or censored at last SD or better.
Time Frame: Baseline up to Cycle 36 (21-day cycles) until disease progression, death or EOT (approximately up to 24.8 months)
Population: Response-Evaluable population includes patients that are either RECIST-evaluable or PSA-evaluable. Here, number of participants analyzed are the participants who were responders. A responder that did not experience disease progression were censored at the last response assessment that is SD or better.
Measure: Median (Full Range); unit: days
Arm/Group | Alisertib 10 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 20 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 + GCSF | Alisertib 40 mg (5D) + Docetaxel 75 mg/m^2 + GCSF
Number analyzed (Participants) | 3 | 1 | 1 | 1 | 0 | 1 | 0 | 1
days | 187 [43 to 187] | 342 [342 to 342] | 830 [830 to 830] | 176 [176 to 176] |  | 79 [79 to 79] |  | NA [1 to 1] — Median values were censored.

14. Secondary Outcome: Duration of Stable Disease (SD)
Description: Duration of SD is defined as the time from first dose to first PD, or censored at last SD or better.
Time Frame: Baseline up to Cycle 36 (21-day cycles) until disease progression, death or EOT (approximately up to 24.8 months)
Population: Response-Evaluable population includes patients that are either RECIST-evaluable or PSA-evaluable. Here, number of participants analyzed are the participants who had SD. For a participants that has not progressed, duration of SD is censored at the last response assessment that is SD or better.
Measure: Median (Full Range); unit: days
Arm/Group | Alisertib 10 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 20 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 + GCSF | Alisertib 40 mg (5D) + Docetaxel 75 mg/m^2 + GCSF
Number analyzed (Participants) | 3 | 6 | 0 | 0 | 1 | 0 | 0 | 1
days | 253 [85 to 253] | NA [169 to 751] — Median values were censored. |  |  | 309 [309 to 309] |  |  | 134 [134 to 134]

ADVERSE EVENTS:
Time Frame: From signing of the informed consent form up to 30 days after the last dose of study drug (up to 25.8 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Alisertib 10 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 20 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 | Alisertib 30 mg (7D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 60 mg/m^2 | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 + GCSF | Alisertib 40 mg (5D) + Docetaxel 75 mg/m^2 + GCSF
Serious Adverse Events (participants affected / at risk) | 3/6 | 10/15 | 3/5 | 2/3 | 1/2 | 3/4 | 2/2 | 2/4
Other Adverse Events (participants affected / at risk) | 6/6 | 14/15 | 5/5 | 3/3 | 2/2 | 4/4 | 2/2 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alisertib 10 mg (7D) + Docetaxel 75 mg/m^2 (N=6) | Alisertib 20 mg (7D) + Docetaxel 75 mg/m^2 (N=15) | Alisertib 30 mg (7D) + Docetaxel 75 mg/m^2 (N=5) | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 (N=3) | Alisertib 30 mg (7D) + Docetaxel 60 mg/m^2 (N=2) | Alisertib 30 mg (5D) + Docetaxel 60 mg/m^2 (N=4) | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 + GCSF (N=2) | Alisertib 40 mg (5D) + Docetaxel 75 mg/m^2 + GCSF (N=4)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 6 | 1 | 1 | 1 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with MLN8237 20 mg + Docetaxel 75 mg/m^2 and is not related to treatment.
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with MLN8237 30 mg (5D) + Docetaxel 75 mg/m^2 and is not related to treatment.
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with MLN8237 30 mg (5D) + Docetaxel 75 mg/m^2 and is not related to treatment.
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alisertib 10 mg (7D) + Docetaxel 75 mg/m^2 (N=6) | Alisertib 20 mg (7D) + Docetaxel 75 mg/m^2 (N=15) | Alisertib 30 mg (7D) + Docetaxel 75 mg/m^2 (N=5) | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 (N=3) | Alisertib 30 mg (7D) + Docetaxel 60 mg/m^2 (N=2) | Alisertib 30 mg (5D) + Docetaxel 60 mg/m^2 (N=4) | Alisertib 30 mg (5D) + Docetaxel 75 mg/m^2 + GCSF (N=2) | Alisertib 40 mg (5D) + Docetaxel 75 mg/m^2 + GCSF (N=4)
Diarrhoea (Gastrointestinal disorders) | 4 | 9 | 1 | 0 | 1 | 1 | 1 | 3
Stomatitis (Gastrointestinal disorders) | 1 | 9 | 2 | 1 | 0 | 1 | 1 | 4
Constipation (Gastrointestinal disorders) | 2 | 4 | 4 | 2 | 0 | 3 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 7 | 2 | 0 | 1 | 2 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 7 | 3 | 0 | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 2 | 0 | 0 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 3 | 0 | 1 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Rectal discharge (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal mass (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 6 | 9 | 5 | 3 | 2 | 4 | 2 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 6 | 3 | 3 | 1 | 3 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 4 | 2 | 1 | 1 | 2 | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 10 | 4 | 1 | 2 | 1 | 2 | 2
Oedema peripheral (General disorders) | 3 | 3 | 1 | 1 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site erythema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site haematoma (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 4 | 5 | 3 | 1 | 2 | 0 | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 4 | 2 | 1 | 0 | 1 | 1 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 5 | 0 | 0 | 2 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 2 | 1 | 0 | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 1 | 5 | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 7 | 3 | 1 | 2 | 1 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 0 | 0 | 0 | 1 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Onychalgia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 4 | 4 | 2 | 1 | 1 | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 5 | 1 | 0 | 0 | 1 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 5 | 0 | 1 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 2 | 0 | 1 | 0 | 2 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatophytosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital infection fungal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 2 | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 0 | 2 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 2 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pallor (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dacryostenosis acquired (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Weight increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urine cytology abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Bladder pain (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oliguria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stoma site pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Device occlusion (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombosis in device (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.